CLINICAL TRIAL: NCT02302196
Title: Autologous Fat Grafting of the Breast in Women With Post Lumpectomy Contour Defects
Status: Completed | Type: Observational
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Other Study IDs: KPNW Fat Grafting 001
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Cancer of the Breast; Anomaly of Breast
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Autologous Fat Grafting of the breast: Approximately 100 women who have had a lumpectomy and qualify, will be offered Autologous Fat Grafting (AFG) procedure. Patients will be assessed 3 months post grafting for safety and efficacy by Breast-Q survey, mammography BIRADS scoring and physical assessment. The AFG may be repeated x 2 at a 3-6 month interval if deemed necessary by the treating surgeon, then reassessed again 3 months later in the same way. Repeat mammogram will be done 1 year post AFG.
  Interventions: Procedure: Autologous Fat Grafting of the Breast
- Control arm standard treatment: Retrospective chart review will be done in 100 women who have undergone standard treatment for breast contour defect after lumpectomy.The control group will be measured by compiling BIRADS scores as well as frequency of subsequent surgical intervention (as necessitated by increased BIRADS scores or by new physical findings on exam) over a 5 year period post lumpectomy.
  Interventions: Other: Control Arm

INTERVENTIONS:
Procedure: Autologous Fat Grafting of the Breast — In fat grafting, fat tissue is removed from other parts of the body; usually thighs, belly, and buttocks by liposuction. The tissue is then processed and injected into the breast area to reconstruct or recreate the breast. The fat will be removed from by a narrow surgical instrument (cannula) through a small incision. Then the fat will be prepared in a specific way before being replaced back in the body. This preparation may include washing, filtering, and centrifugation (spinning) of the fat. The fat is then placed into the desired area of the breast using either a smaller cannula or needle.
  Groups: Autologous Fat Grafting of the breast
Other: Control Arm — Retrospective chart review for women who have undergone standard breast reconstruction for lumpectomy.
  Groups: Control arm standard treatment

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of breast reconstruction using Autologous Fat Grafting (AFG) for women post lumpectomy that have contour defects.

The study hypothesis is that AFG has emerged as a less invasive alternative to breast reconstruction post mastectomy. AFG could be used to treat breast contour defects with much less invasive outpatient surgery, using the patient's own cells and tissues, which overall reduces risk.

DETAILED DESCRIPTION:
About 200 women at Kaiser Permanente Northwest will be in this study. The study will include about 100 women who have had a lumpectomy and consent to be in the research arm and have AFG and 100 from the control arm (retrospective chart review).

Autologous Fat Grafting Arm: Breast-Q survey of patient satisfaction will be collected before and after AFG. Assessments will be done 3 months post grafting for efficacy (excellent 100% correction of defect), good (75% correction of defect), fair (50% correction of defect), poor 25% or less correction of defect) result will be recorded. AFG may be repeated x 2 at a 3-6 month interval if deemed necessary by the treating surgeon, then reassessed again 3 months later in the same way. A mammographic assessment of the breast, scored by radiologist in a 6 step scoring system (BIRADS score) will be done 1 year after AFG. BIRADS scores and new physical finding will continue to be collected for a 5 year period post AFG post lumpectomy group.

Control (non-Autologous Fat Grafting) arm: Retrospective chart review for women who have undergone standard treatment to treatment to reconstruct their breasts. Data collected will include; BIRADS scores as well as frequency of subsequent surgical intervention (as necessitated by increased BIRADS scores or by new physical findings on exam) over a 5 year period post lumpectomy.

.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age 18 > y/o
* If patient has had lumpectomy and radiation, need to be at least 3 years out from completion of radiation
* Must be a Kaiser Permanente Northwest Member

Exclusion Criteria:

* Active smokers, cannot quit smoking for at least one month before and after procedures
* Patients who have such extensive skin scarring that elasticity is lost
* Patients who have little to no subcutaneous donor fat
* Patients with BIRAD's 3 or greater mammograms after treatment
* Patients with aggressive cancer for which cure is the goal (do not want to exclude patients that want palliative procedure) - inflammatory breast cancer
* Patients with triple negative cancer - ER -, PR -, Her2-neu -
* Patients with BRCA or CHEK-2 gene mutations or those with strong family history of breast cancer [more than 2 first degree relatives with breast cancer]
* Patients that have had a lumpectomy for breast cancer who have declined radiation therapy when it was recommended to reduce risk of local recurrence (should not exclude patients over 70 y/o who have elected to have lumpectomy and anti-estrogen therapy instead of lumpectomy and radiation)
* Oncoplastic reduction patients
* Comorbidities that preclude multiple procedures being done
* Pregnant women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kaiser Permanente Northwest members (women) who have undergone lumpectomy and radiation treatment.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2015-09; Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Safety of Autologous Fat Grafting (AFG) compared to standard breast reconstruction for lumpectomy, as measured by the BIRADS scores | 5 years for lumpectomy
  The experimental AFG group will have the same or less change in the BIRADS scores than the control non-AFG group.

SECONDARY OUTCOMES:
Women undergoing Autologous Fat (AFG) Grafting of the breast | Prior to AFG and 1 year after procedure
  The Breast Q survey will be administered to women before and after the AFG procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Murphy, MD, Principal Investigator — Kaiser Permanente Northwest Region
Locations (1):
- Kaiser Permanente NW Region, Sunnybrook Medical Office Building, Clackamas, Oregon, United States

IPD SHARING:
Plan to Share IPD: No